CLINICAL TRIAL: NCT05578794
Title: The Effect of Straining Techniques on Duration of Labor, Perineal Trauma Status, and Newborn Apgar Score
Brief Title: The Effect of Straining Techniques on Women and Newborn
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Ozlem Akgün, Lecturer, Cumhuriyet University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: OAkgun
Record Dates: First submitted 2022-10-05; First posted 2022-10-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Prolonged Second Stage of Labor; Other Specified Trauma to Perineum and Vulva During Delivery; Newborn; Vitality
Keywords: Labor; Midwife; Pregnant; Straining techniques; Perineal trauma; Apgar Score

STUDY DESIGN:
Intervention Model Description: Valsalva-type Straining (Group I), Spontaneous Straining (Group II), Natural Straining (Group III))
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Valsalva Straining (Control Group) (Experimental): The straining techniques for the groups were explained by the researcher in line with the process steps in the latent phase. Valsalva straining is supported in 2nd stage of labor. Duration of delivery, perineal trauma status and Apgar Scores were evaluated.
  Interventions: Other: Straining types
- Spontaneous Straining (Experimental): The straining techniques for the groups were explained by the researcher in line with the process steps in the latent phase. Spontaneous straining is supported in 2nd stage of labor. Duration of delivery, perineal trauma status and Apgar Scores were evaluated.
  Interventions: Other: Straining types
- Natural Straining (Experimental): The straining techniques for the groups were explained by the researcher in line with the process steps in the latent phase. Duration of delivery, perineal trauma status and Apgar Scores were evaluated.
  Interventions: Other: Straining types

INTERVENTIONS:
Other: Straining types — Valsalva, spontaneous and natural strainings are supported in 2nd stage of labor. Duration of delivery, perineal trauma status and Apgar Scores were evaluated.

SUMMARY:
Purpose: To examine the effects of straining techniques on the duration of labor, perineal trauma status and newborn apgar score.

Method: This study is a randomized controlled trial. The straining techniques were explained to the pregnant women who gave written consent to participate in the study and were randomly assigned to groups in the latent phase (natural, spontaneous, Valsalva), and the techniques were applied in the second phase of labor.

DETAILED DESCRIPTION:
Purpose: The present study was planned to determine the effects of straining techniques on the duration of labor, perineal trauma status, and newborn Apgar score.

Method: The study, which had a randomized-controlled experimental design, was conducted in Sivas Numune Hospital Birth Unit. The sampling size was calculated using power analysis. In the literature, spontaneous straining is used by pregnant women in the range of 25-81%, and Valsalva -type straining has a rate of 32-75%. To represent the population of the study, sample volume was determined at =0.05 significance level, 1- =0.95 Confidence Interval, =0.20 error risk, and 1- =0.80 power, and the total number of individuals was determined as 354. The data of the study were collected with the "Pre-Evaluation Form", "Personal Information Form", "Labor Evaluation Form", and "Apgar Score" created by the researchers in line with the literature data. The straining techniques were explained to the pregnant women who gave written consent to participate in the study and were randomly assigned to groups in the latent phase (natural, spontaneous, Valsalva), and the techniques were applied in the second phase of labor. ANOVA, Kruskal Wallis H-test, Chi-square test, Exact test, Tamhane T2 test, and Dunn Test were used to evaluate the data obtained in the study. Statistical significance was evaluated at a 0.05 significance level and the SPSS version 23.0 was used.

ELIGIBILITY:
Inclusion Criteria:

* 38-42. being at the gestational week,
* Having a singleton pregnancy
* Fetus in vertex position
* Being in the latent phase in the first stage of labor
* Planning and having a normal vaginal birth,
* Not having a diagnosed chronic physical disease,
* Not having a diagnosed psychiatric disease,
* No risk of risky pregnancy or fetal anomaly,
* Being literate,
* No communication problem
* Giving birth in the lithotomy position
* Volunteering to participate in the study

Exclusion Criteria:

* 38-42. not in the week of pregnancy,
* Having multiple pregnancy
* Fetus out of vertex position
* Being in the latent phase in the first stage of birth,
* Having a cesarean section while planning a normal vaginal delivery,
* Having a diagnosed chronic physical illness,
* Having a diagnosed psychiatric illness,
* Having a risky pregnancy or fetal anomaly risk,
* illiteracy,
* Having a communication problem
* Giving birth in different positions
* Not willing to participate in the study

Ages: 19 Years to 41 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 354 (Actual)
Dates: Start 2020-02-24 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
The distribution of the duration of the second phase according to the straining styles of women in labor | 2-90 minute
  The distribution of the duration of the second phase was evaluated according to the pushing styles of the women who gave birth. The duration of the second stage of labor was calculated by keeping the hours and minutes according to the type of straining used. The time from the woman's full dilation (10 cm) to the birth of the baby was measured.
The perineal trauma status according to the straining styles of women during labor | 10-30 minute
  Perineal trauma status of women was evaluated according to their pushing styles during delivery. Episiotomy or laceration status after delivery of the placenta was evaluated by observation and examination method.
The distribution of the mean Apgar Scores of the newborns according to the straining types of women during labor | 1-5 minute
  The newborn apgar scores were evaluated according to the straining types of the women at the time of delivery. Apgar Score is the expression of the physiological condition of the infant at a certain time (ACOG, 2015). In studies examining the relationship between mortality rates and Apgar scores, it was shown that infants with low scores (0-2) had higher mortality rates (14%). Infants with high scores (7-10) had lower mortality rates (0.13%). The scoring system showed that overall Apgar scores of infants born with cesarean section were lower than those born vaginally (Apgar, 1966; Rubarth, 2012). Apgar developed this evaluation tool with 5 objective criteria (heart rate, respiration, reflex irritability, muscle tonus, and color). The Apgar Evaluation System is used in the 1st and 5th minutes after the infant is born. Apgar scores of 7-10 are reassuring, normal, 4-6 moderately abnormal, and 0-3 are considered low in term and preterm infants (ACOG, 2015).

SECONDARY OUTCOMES:
The distribution of women's satisfaction and considerations about the practice according to the way they strain during labor | 30 minute- 4 hours
  According to the types of straining during childbirth, women's satisfaction and thoughts about the application were evaluated. The satisfaction of women with the pushing techniques was evaluated with the questions asked in the questionnaire. Each woman was asked whether she would like to use the type of pushing she used in her next birth.

CONTACTS AND LOCATIONS:
Overall Officials: Gulbahtiyar Demirel, Principal Investigator — Cumhuriyet University
Locations (1):
- Sivas sample hospital, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Second Stage of Labor — http://doi.org/10.1097/GRF.0000000000000113
- See also: Is directed open-glottis pushing more effective than directed closed-glottis pushing during the second stage of labor? A pragmatic randomized trial-the EOLE study. — http://doi.org/10.1016/j.midw.2020.102843
- See also: The impact of valsalva's versus spontaneous pushing techniques during second stage of labor on postpartum maternal fatigue and neonatal outcome. — http://www.sjmms.net/text.asp?2014/2/2/101/137000